CLINICAL TRIAL: NCT01606839
Title: Noninvasive Measurement of Cardiac Output in Pulmonary Hypertension Using Inert Gas Rebreathing
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Collaborators: Ludwig Boltzmann Gesellschaft (Other)
Responsible Party: Sponsor
Other Study IDs: 24-079 ex 11/12
Record Dates: First submitted 2012-05-24; First posted 2012-05-28 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study hypothesis is that accuracy of CO measurement by IGR does not differ from classical CO measurement methods such as thermodilution or direct Fick method. This is why the study aims to determine whether non invasive cardiac output (CO) measurement using inert gas rebreathing (IGR)is a suitable method in patients with pulmonary hypertension. In order to examine this, the IGR method will be used in patients undergoing diagnostic or follow-up right heart catheterization.

DETAILED DESCRIPTION:
Inert Gas Rebreathing method enables non invasive measurement of cardiac output (CO) using the single rebreathing method. A mixture of blood soluble (N2O) and blood insoluble gas (SF6) and environmental air is inhaled and the amount of N2O, SF6, O2 and CO2 is measured by a photoacoustic analysator. The length of a measurement is about 1 minute.

As the gold standard measurement of CO is performed invasively, there is an urgent need for the development of non-invasive tools like IGR.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Patients who undergo right heart catheterization

Exclusion Criteria:

* Missing written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients undergoing diagnostic or follow-up right heart cathereization.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2012-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Cardiac output | at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Horst Olschewski, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Ludwig Boltzmann Institute for Lung Vascular Research, Graz, Austria